CLINICAL TRIAL: NCT06754267
Title: Venetoclax Combined With Olverembatinib and Predinisone in Treating Ph-positive Precursor B Cell Acute Lymphoblastic Leukemia: a Phase II, Single Arm and Multicenter Study
Brief Title: Venetoclax Combined With Olverembatinib and Predinisone in Treating Ph+ B-ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT20240094C
Record Dates: First submitted 2024-12-18; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Precursor B-Cell Acute Lymphoblastic Leukemia
Keywords: acute lymphoblastic leukemia; Ph chromosome; BCL2 inhibitor; TKI
MeSH Terms: conditions — Precursor B-Cell Lymphoblastic Leukemia-Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — venetoclax; olverembatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): Induction Cycle 1: Olverembatinib for 4 weeks, oral; Venetoclax for 4 weeks, oral; Predinisone for 3 weeks, oral.
  Consolidation Cycle 2 and 3: Olverembatinib for 4 weeks, oral; Venetoclax for 2 weeks, oral; Predinisone for 2 weeks, oral.
  Interventions: Drug: Venetoclax; Drug: Olverembatinib; Drug: Predinisone

INTERVENTIONS:
Drug: Venetoclax — BCL-2 inhibotor
  Other Names: Ven
Drug: Olverembatinib — Tyrosine kinase inhibitor
  Other Names: Olv
Drug: Predinisone — Glucocorticoids

SUMMARY:
Precursor B cell acute lymphoblastic leukemia (B-ALL) is an aggressive type of leukemia, with high relapse rate and poor long term survival in adults. Philadelphia chromosome positive (Ph+) ALL is defined as ALL with translocation between chromosomes 9 and 22. And t(9;22)(q34;q11) is the most common chromosomal abnormality in ALL. Before the emergence of TKI, the prognosis of Ph+ ALL was extremely poor, and the long-term survival rate was only 10%-35%. Ph+ ALL accounts for about 30% of adult ALL. In this study, the investigators propose a treatment approach that combines Venetoclax with Olverembatinib and Predinisone in Ph+ B-ALL adults. The study aims to answer the safety and efficacy of this treatment regimen, and further improve the survival for those participants.

DETAILED DESCRIPTION:
This is a prospective, single-arm, phase II and open-label study. A total of 36 Ph-positive B-ALL participants will be enrolled. The primary endpoint is complete molecular response (CMR) after three cycles of venetoclax combined with olverembatinib and prednisone regimen (VOP) in the treatment of de novo acute Philadelphia chromosome-positive (Ph+) B-lymphoblastic leukemia. The purpose of this study is to explore the safety and efficacy of the multi-drug combination regimen in the treatment of newly diagnosed Ph-positive B-ALL patients.

ELIGIBILITY:
Inclusion Criteria:

1. Before enrollment, the patient must be diagnosed with de novo precursor B-cell acute lymphoblastic leukemia and positive for Philadelphia chromosome (presence of t(9;22) and/or BCR::ABL1 positive and/or FISH positive). The diagnostic criteria refer to the 2022 WHO classification;
2. Age ≥ 18 years;
3. Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2;
4. Expected survival time ≥ 3 months;
5. No organ dysfunction that would restrict the use of this protocol during the screening period;
6. Understand the study and sign the informed consent form.
7. Men, women of childbearing age (only postmenopausal women who have been menopausal for at least 12 months can be considered infertile), and their partners voluntarily take effective contraceptive measures deemed effective by the investigator during the treatment period and for at least 12 months after the last dose of the study drug.

Exclusion Criteria:

1. Accelerated phase or blast crisis of chronic myeloid leukemia;
2. Subjects with involvement of the central nervous system (CNS) or accompanied by extramedullary lesions;
3. Subjects who have received systemic anti-leukemia treatment (including but not limited to TKI, radiotherapy or chemotherapy, except for the allowed pretreatment);
4. Subjects with a history of myocardial infarction within 12 months, or have clinical manifestations of heart disease (including but not limited to unstable angina pectoris, congestive heart failure, uncontrolled hypertension and uncontrolled arrhythmia, etc.); left ventricular ejection fraction (LVEF) on echocardiography <50%;
5. Diseases with abnormal functions of organs such as lung, liver, and kidney that may limit the patient's participation in this trial (including but not limited to severe infection, uncontrolled diabetes, active tuberculosis, asthma, COPD, bronchiectasis, etc.);
6. History of other malignancies within the past 5 years, excluding localized thyroid cancer and in situ skin cancer;
7. Serum total bilirubin > 1.5 ULN (upper limit of normal); ALT or AST > 2.5 ULN; serum creatinine > 1.5 ULN;
8. Known HIV infection;
9. Conditions affecting the use of the study drug as assessed by the investigator;
10. Unable to understand or comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
complete molecular response (CMR) after three cycles | At the end of Cycle 3（each cycle is 28 days）
  BCR::ABL1≤0.01% detected by RT-qPCR

SECONDARY OUTCOMES:
Complete remission with or without incomplete PB cell recovery(CR/CRi) rate | after Cycle 1(each cycle is 28 days)
  Blast rate lower than 5% with or without peripheral blood cell recover
Event free survival (EFS) | up to 2 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first;
Overall survival (OS) | up to 2 years
  Defined for all patients in a trial; measured from day 1 of treatment to the date of death from any cause;
Minimal residual disease (MRD) | At the end of each cycle（each cycle is 28 days）, up to 2 years
  MRD level detected by flow cytometry which value <0.1% is defined as negtive; MRD level detected by RT-qPCR which BCR::ABL1 value <0.01% is defined as negtive
Relapse free survival(RFS) | up to 2 years
  Defined only for patients achieving CR or CRi; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause;
Incidence of Adverse Events | From day 1 of treatment to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.Hematologic and non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravandi F, Jorgensen JL, Thomas DA, O'Brien S, Garris R, Faderl S, Huang X, Wen S, Burger JA, Ferrajoli A, Kebriaei P, Champlin RE, Estrov Z, Challagundla P, Wang SA, Luthra R, Cortes JE, Kantarjian HM. Detection of MRD may predict the outcome of patients with Philadelphia chromosome-positive ALL treated with tyrosine kinase inhibitors plus chemotherapy. Blood. 2013 Aug 15;122(7):1214-21. doi: 10.1182/blood-2012-11-466482. Epub 2013 Jul 8. PMID 23836561
- [Background] Kim DY, Joo YD, Lim SN, Kim SD, Lee JH, Lee JH, Kim DH, Kim K, Jung CW, Kim I, Yoon SS, Park S, Ahn JS, Yang DH, Lee JJ, Lee HS, Kim YS, Mun YC, Kim H, Park JH, Moon JH, Sohn SK, Lee SM, Lee WS, Kim KH, Won JH, Hyun MS, Park J, Lee JH, Shin HJ, Chung JS, Lee H, Eom HS, Lee GW, Cho YU, Jang S, Park CJ, Chi HS, Lee KH; Adult Acute Lymphoblastic Leukemia Working Party of the Korean Society of Hematology. Nilotinib combined with multiagent chemotherapy for newly diagnosed Philadelphia-positive acute lymphoblastic leukemia. Blood. 2015 Aug 6;126(6):746-56. doi: 10.1182/blood-2015-03-636548. Epub 2015 Jun 11. PMID 26065651
- [Background] Sasaki K, Kantarjian HM, Short NJ, Samra B, Khoury JD, Kanagal Shamanna R, Konopleva M, Jain N, DiNardo CD, Khouri R, Garcia-Manero G, Kadia TM, Wierda WG, Khouri IF, Kebriaei P, Mehta RS, Champlin RE, Garris R, Cheung CM, Daver N, Thompson PA, Yilmaz M, Ravandi F, Jabbour E. Prognostic factors for progression in patients with Philadelphia chromosome-positive acute lymphoblastic leukemia in complete molecular response within 3 months of therapy with tyrosine kinase inhibitors. Cancer. 2021 Aug 1;127(15):2648-2656. doi: 10.1002/cncr.33529. Epub 2021 Apr 1. PMID 33793964
- [Background] Tang H, Jia W, Jia S, Dong R, Gao S, Feng J, Dong H, Gu H, Zhang T, Yuan R, Liu X, Cheng L, Zhou S, Gao G. A new chemotherapy-free regimen of olverembatinib in combination with venetoclax and dexamethasone for newly diagnosed Ph+ acute lymphoblastic leukemia: Preliminary outcomes of a prospective study. Am J Hematol. 2024 Jun;99(6):1177-1179. doi: 10.1002/ajh.27289. Epub 2024 Mar 14. No abstract available. PMID 38482543
- [Background] Ravandi F, O'Brien SM, Cortes JE, Thomas DM, Garris R, Faderl S, Burger JA, Rytting ME, Ferrajoli A, Wierda WG, Verstovsek S, Champlin R, Kebriaei P, McCue DA, Huang X, Jabbour E, Garcia-Manero G, Estrov Z, Kantarjian HM. Long-term follow-up of a phase 2 study of chemotherapy plus dasatinib for the initial treatment of patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Cancer. 2015 Dec 1;121(23):4158-64. doi: 10.1002/cncr.29646. Epub 2015 Aug 26. PMID 26308885
- [Background] Daver N, Thomas D, Ravandi F, Cortes J, Garris R, Jabbour E, Garcia-Manero G, Borthakur G, Kadia T, Rytting M, Konopleva M, Kantarjian H, O'Brien S. Final report of a phase II study of imatinib mesylate with hyper-CVAD for the front-line treatment of adult patients with Philadelphia chromosome-positive acute lymphoblastic leukemia. Haematologica. 2015 May;100(5):653-61. doi: 10.3324/haematol.2014.118588. Epub 2015 Feb 14. PMID 25682595
- [Background] Fielding AK, Rowe JM, Buck G, Foroni L, Gerrard G, Litzow MR, Lazarus H, Luger SM, Marks DI, McMillan AK, Moorman AV, Patel B, Paietta E, Tallman MS, Goldstone AH. UKALLXII/ECOG2993: addition of imatinib to a standard treatment regimen enhances long-term outcomes in Philadelphia positive acute lymphoblastic leukemia. Blood. 2014 Feb 6;123(6):843-50. doi: 10.1182/blood-2013-09-529008. Epub 2013 Nov 25. PMID 24277073
- [Background] Groffen J, Stephenson JR, Heisterkamp N, de Klein A, Bartram CR, Grosveld G. Philadelphia chromosomal breakpoints are clustered within a limited region, bcr, on chromosome 22. Cell. 1984 Jan;36(1):93-9. doi: 10.1016/0092-8674(84)90077-1. PMID 6319012
- [Background] NOWELL PC, HUNGERFORD DA. Chromosome studies on normal and leukemic human leukocytes. J Natl Cancer Inst. 1960 Jul;25:85-109. No abstract available. PMID 14427847